CLINICAL TRIAL: NCT07379359
Title: The ADHD Kids´ Study: Randomized Clinical Trial on the OutSMARTers Program and Individual Counseling for Children Aged 9-12 With ADHD
Brief Title: The ADHD Kids´ Study for Children 9-12 Years of Age
Acronym: OutSmarters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Principal Investigator, Dagmar Kristín Hannesdóttir, Assistant professor, Department of Psychology, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI-2025-OutSMARTersADHDstudy; 94059 (Other Grant/Funding Number: University of Iceland Research Fund)
Record Dates: First submitted 2025-09-27; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: Intervention program for ADHD; Children; OutSMARTers Program; Skill building; Cognitive-behavioral therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The proposed study is an RCT with a three-group parallel design. The children will be randomly assigned to three groups using a 2:2:1 ratio: 1) The OutSMARTers program (n = 40), 2) The Kid Counseling Program (n = 40) or 3) A wait-list control group (n = 20), which will receive the OutSMARTers program or the Kid Counseling Program once the waiting period (5 weeks) is over.
Masking Description: Teachers of the enrolled children will be completing assessments before and after the interventions and will be blind to the treatment / wait list allocation of the child they are reporting on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The OutSMARTers program (Experimental): Child directed group skills training and cognitive-behavior therapy
  Interventions: Behavioral: The OutSMARTers Program
- The Kid Counseling Program (Experimental): Child directed individual sessions, skills training and cognitive-behavior therapy.
  Interventions: Behavioral: The Kid Counseling Program
- Wait-list control group (No Intervention): The Wait-list control group is assessed at pre and post (five week interval) and then receives either the OutSMARTers program or the Kid Counseling Program.

INTERVENTIONS:
Behavioral: The OutSMARTers Program — An intervention specifically designed to improve common difficulties that children with ADHD wrestle with daily. The program consists of ten sessions (90 minutes each) conducted by two or three trainers working with a group of six children over the course of five weeks. The children attend four different stations during the intervention: the Emotion station and the Friendship station in sessions one through five, and the Stopping station and the Solution station in the remaining five. The program is fully manualized and was published in Icelandic in 2017 (Hannesdottir et al., 2017b). A small RCT pilot study of the OutSMARTers program delivered in a clinical setting showed beneficial effects on emotion regulation skills, social skills and a reduction in ADHD symptoms as rated by parents (Hannesdottir et al., 2017a).
  Arms: The OutSMARTers program
Behavioral: The Kid Counseling Program — The Kid Counseling Program consists of five 50-minute individual counseling sessions, each delivered by a professional, and based on the book Learning to Slow Down and Pay Attention (Nadeau & Dixon, 2004). The content closely mirrors that of the OutSMARTers program and shares the same goal; to improve common deficits that children with ADHD face. The key difference is that, unlike the OutSMARTers program, this intervention is individualized and does not include peer-based practice of the skills learned.
  Arms: The Kid Counseling Program

SUMMARY:
The aim of the study is to compare the efficacy of The OutSMARTers program- an ADHD skills training group program for children aged 9-12 to customized individual counseling provided by a professional, The Kid Counseling Program. Approximately 100 children will be randomly assigned to either intervention or a small wait-list group who will after a five-week-waiting period receive either intervention. Following the intervention, parents, children, and teachers will evaluate the effects on communication skills, well-being, and emotional regulation.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is an impairing neurodevelopmental disorder among children and adolescents that makes it difficult to cope with challenges of everyday life. Although various interventions have been developed to support parents of children with ADHD, few have been specifically designed for the children themselves, particularly interventions that focus directly on emotion regulation, problem-solving, communication and emotional well-being. The study is a randomized controlled trial (RCT) comparing the effectiveness of the OutSMARTers program, a skills-training group program based on cognitive- behavioral therapy (CBT) elements for children with ADHD. The program includes training in emotional regulation, social skills, self-control and problem-solving within a behavior modification framework. The comparison intervention, The Kid Counseling Program, consists of five sessions of individual counseling with similar content as in the OutSMARTers program, provided by a professional. The participants of this study will be approximately 100 children aged 9-12 that have been diagnosed with ADHD. Various methods will be used to assess outcomes, drawing on data from multiple sources through repeated measurements, including reports from parents, teachers, and the children themselves. The scientific goal of the study is to evaluate the efficacy of the OutSMARTers program, a group- based intervention delivered in 10 sessions over the course of 5 weeks, compared to brief individual counseling provided by a professional but not in a group of same-age peers. Positive changes in emotional regulation, communication skills, and well-being are expected in both groups. However, it is also possible that certain subgroups (e.g. children with or without comorbidities such as anxiety) may benefit more from one intervention over the other.

ELIGIBILITY:
Inclusion Criteria:

* age: 9-12
* have an ADHD diagnosis confirmed by a school psychologist
* children need to be fluent in Icelandic
* Parents need to be fluent in Icelandic or English

Exclusion Criteria:

* Children need to have an IQ of 70 or higher (WISC-IV test or WPSSI-R test)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Strengths and difficulties questionnaire (SDQ) | Baseline, upon completion of 5 week program, at the 6 month follow-up
  SDQ assess behavior and well-being in children generally based on the following factors: emotional problems, behavioral problems, hyperactivity, social difficulties, and social competence. Each item is scored on a 0-2-point Likert scale, where higher scores indicate more difficulties, except on the social competence factor. Higher scores on the social competence factor indicate better social competence.
Emotion Regulation Checklist (ERC) | Baseline, upon completion of 5 week program, 6 month follow-up
  The ERC measures emotion regulation among youth. Parents and teachers complete this questionnaire regarding the child's emotional regulation and negative mood. The scale consists of 24 questions and has been validated in the general Icelandic population. Each item is scored on a 1-4 Likert Scale. Higher scores on the Lability/Negativity factor indicate more dysregulation and difficulties. while higher scores on the Emotion Regulation factor indicate better emotion regulation skills.
ADHD Rating Scale (ADHD) | Baseline, upon completion of 5 week program, 6 month follow-up
  The ADHD scale assesses symptoms and impairment of attention-deficit/hyperactivity disorder, i.e. difficulties with concentration and hyperactive behavior. These symptoms align with the diagnostic criteria of the DSM classification system. Each item is scored on a 0-3 Likert Scale where higher scores indicate more ADHD symptoms. Responses from parents and teachers are compared to the norms of Icelandic children.
Revised Children's Anxiety and Depression Scale (RCADS) | Baseline, upon completion of 5 week program, 6 month follow-up
  The RCADS is a commonly used questionnaire to screen for anxiety and depressive disorders and to assess changes following an intervention. The RCADS is a 47-item questionnaire designed for parents and children (ages 8-17) and includes the following scales: Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Obsessive-Compulsive Disorder, and Depressive Symptoms. Items are rated on a four-point scale: 0 = never, 1 = sometimes, 2 = often, 3 = always. Higher scores indicate more anxiety and depressive symptoms. The Icelandic version has acceptable psychometric properties in both general and clinical populations.
Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents-Revised Version (KINDL-R) | Baseline, upon completion of 5 week program, 6 month follow-up
  Parents and children are asked to evaluate how well the child has been doing and feeling recently in terms of physical health, emotional well-being, self-esteem, family relationships, peer relationships, and school (Ravens-Sieberer & Bullinger, 1998 - see www.kindl.org). Each item is scores on a Likert scale of 1-5 and higher scores indicate better quality of life for each factor.
Social Skills Rating System (SSRS) | Baseline, upon completion of 5 week program, 6 month follow-up
  Children complete an assessment on their social skills. The questionnaire assesses Cooperation, Assertion, Self-control and Responsibility. Items are scored on a 0-2 Likert scale where higher scores on each factor indicates better skills.
Treatment satisfaction | Upon completion of 5 week program
  Parents and children complete questions on treatment satisfaction. The questions include some open comments, but most items are scored on a scale of 1-4, with higher ratings indicating more satisfaction.

IPD SHARING:
Plan to Share IPD: No
As the study includes repeated measures of a clinical child population, parts of the data will be classified as sensitive personal data and thus restricted by the permit from the National Bioethics Committee of Iceland.

REFERENCES:
- [Background] Hannesdottir DK, Ingvarsdottir E, Bjornsson A. The OutSMARTers Program for Children With ADHD. J Atten Disord. 2017 Feb;21(4):353-364. doi: 10.1177/1087054713520617. Epub 2016 Jul 28. PMID 24505061